CLINICAL TRIAL: NCT04547244
Title: Optimization of Cardiac Resynchronization Therapy and Its Effects in Patients With Type 2 Diabetes Mellitus: Automatic Optimization vs. Echocardiographic Guided Optimization.
Brief Title: CRTd Responders Optimization
Status: Completed | Type: Observational
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Celestino Sardu, researcher, University of Campania Luigi Vanvitelli
Other Study IDs: 08.09.20
Record Dates: First submitted 2020-09-07; First posted 2020-09-14 (Actual); Last update posted 2020-09-14 (Actual); Status verified 2020-09

CONDITIONS: Heart Failure; Heart Failure With Reduced Ejection Fraction; Cardiac Death
MeSH Terms: conditions — Heart Failure; Death

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- T2DM patients with CRTd with automatic optimization: In this cohort the T2DM patients with CRTd will receive at follow-up an automatic optimization of CRTd.
- T2DM patients with CRTd with echocardiographic optimization: In this cohort the T2DM patients with CRTd will receive at follow-up an echocardiography guided optimization of CRTd.
  Interventions: Other: echocardiographic optimization of CRTd

INTERVENTIONS:
Other: echocardiographic optimization of CRTd — the patients after the implant of CRTd and during the follow-up will receive an echocardiography to optimize the atrio-ventricular and inter-ventricular delay, and to improve the effects of CRTd.
  Groups: T2DM patients with CRTd with echocardiographic optimization

SUMMARY:
Suboptimal optimization of atrio-ventricular (AV) and inter-ventricular (VV) timings could affect the clinical response of CRTd in T2DM patients. Thus, authors hypothesize that automatic sensor guided CRTd optimization could ameliorate clinical outcomes in patients with T2DM. However, authors will evaluate the effects of cardiac resynchronization therapy (CRTd) in patients with type 2 diabetes mellitus (T2DM) optimized via automatic vs. echocardiographic guided approach.Authors will conduct a prospective, multicenter study to recruit, from October 2016 to June 2019, patients with T2DM and heart failure (HF) candidate to receive a CRTd. After CRTd the patients will be optimized via automatic vs. echocardiographic guided approach.

ELIGIBILITY:
Inclusion Criteria:

* heart failure with reduced cardiac pump, NYHA class II/III, indication to receive a CRTd.

Exclusion Criteria:

* NYHA class IV, previous CRTD implantation, neoplastic disease, inflammatory chronic disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged more than 18 and less than 75 affected by chronic heart failure in NYHA class II/III with reduced cardiac pump and indication to receive a CRTd.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
CRTd responders rate | 12 months
  The authors will evaluate the CRTd responders rate in terms of patients that will experience the reduction of NYHA class, improvement of HF symptoms, and improvement of left ventricle ejection fraction.

CONTACTS AND LOCATIONS:
Locations (1):
- Celestino Sardu, Napoli, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sardu C, Paolisso P, Ducceschi V, Santamaria M, Sacra C, Massetti M, Ruocco A, Marfella R. Cardiac resynchronization therapy and its effects in patients with type 2 DIAbetes mellitus OPTimized in automatic vs. echo guided approach. Data from the DIA-OPTA investigators. Cardiovasc Diabetol. 2020 Nov 28;19(1):202. doi: 10.1186/s12933-020-01180-8. PMID 33248462